CLINICAL TRIAL: NCT05974358
Title: KONO-S Anastomosis Compared to Conventional Ileocolonic Anastomosis to Reduce Recurrence in Crohn's Disease: a Superiority Phase III Prospective, Randomized, Multicenter, Double-blind Trial.
Brief Title: KONO-S Anastomosis Compared to Conventional Ileocolonic Anastomosis to Reduce Recurrence in Crohn's Disease
Acronym: KOALA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023/802
Record Dates: First submitted 2023-07-26; First posted 2023-08-03 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Crohn Disease
Keywords: Crohn's disease; Kono-S anastomosis; conventional anastomosis; endoscopic recurrence
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Intervention Model Description: prospective, multicenter,randomized study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kono-S group (Experimental): Kono-S group, in which ileocolonic anastomosis will be performed following the technique described by Kono et al.
  Interventions: Procedure: Kono-S anastomosis
- Control group (Other): Conventional side-to-side ileocolonic anastomosis
  Interventions: Procedure: Conventional anastomosis for ileocolonicresection of Crohn's disease

INTERVENTIONS:
Procedure: Kono-S anastomosis — Kono et al. described a new operative technique that could reduce the rate of post-operative recurrence: a termino-terminal ileocolonic anastomosis, anti-mesenteric, with a supporting column to prevent distortion and anastomotic stenosis (Kono-S anastomosis).
  Arms: Kono-S group
Procedure: Conventional anastomosis for ileocolonicresection of Crohn's disease — conventional anastomosis for ileocolonicresection of Crohn's disease
  Arms: Control group

SUMMARY:
Crohn's disease (CD) is a chronic inflammatory bowel disease (IBD) currently affecting one person in a thousand in France. It can lead to numerous digestive complications such as fistulas, abscesses or stenosis. Despite numerous therapeutic advances, the rate of patients requiring surgery remains very high, with approximately 50% requiring at least one surgical intervention at 10 years after disease diagnosis. However, surgical treatment is not curative, the postoperative recurrence rate being very high, from 65 to-90% endoscopic recurrence at 1 year. The ileocolonic anastomosis is the main site of postoperative recurrence currently defined by a Rutgeerts score (≥i2) 6 months after surgery. In 2003, Kono et al. described a new operative technique that could reduce the rate of post-operative recurrence: a termino-terminal ileocolonic anastomosis, anti-mesenteric, with a supporting column to prevent distortion and anastomotic stenosis (Kono-S anastomosis). The study showed no decrease in endoscopic recurrence rate at 1 year (83% vs 79%), but a significant decrease in surgical recurrence rate at 5 years (15% vs 0%). Recently, a randomized Italian monocenter study showed a significant decrease in endoscopic recurrence rate at 6 and 18 months (22.2% versus 62.8% and 25% versus 67.4%), as well as a decrease in clinical recurrence. The limitations of this study are its monocentric nature and the lack of centralization of the endoscopic analysis to assess the primary endpoint. This surgical technique has been performed in some centers for ileocolonic Crohn's surgery since 2020. Nevertheless, the level of evidence remains too low to establish practice recommendations. The KOALA study will be the first prospective, multicenter, randomized study comparing KONO-S anastomosis and conventional anastomosis for ileocolonicresection of Crohn's disease, with blinded and centralized evaluation of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ≥ 18 years and ≤75 years
* With Crohn's disease.
* Requiring a first ileocolonic resection: fistulizing, abscessed, or stenosing disease or disease refractory to medical treatment.
* Affiliated to the French social security system.

Exclusion Criteria:

* Previous ileocolonic resection
* Contraindication to postoperative endoscopy.
* Anastomosis with a planned defunctioning protective stoma.
* Emergency surgery (peritonitis).
* Lack of consent to the study.
* Pregnant patients.
* Refusal to participate or inability to provide informed consent.
* Patient under legal protection (individuals under guardianship by court order)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
endoscopy score | Month 6
  Rutgeerts endoscopy score ≥ i2 (>5 anastomotic lesions with passable stenosis (skip lesions); or lesions in the area of the anastomosis) at 6 months obtained by centralized double reading of filmed endoscopy.
  I0 no lesions
  * 1 <5 aphthous lesions in the neoterminal ileum
  * 2 >5 anastomotic lesions with passable stenosis (skip lesions); or lesions in the area of the anastomosis
  * 3 diffuse ileitis
  * 4 diffuse ileitis with deep ulcerations and/or Stenosis

SECONDARY OUTCOMES:
Harvey-Bradshaw Index (HBI) | Month 6
  Harvey-Bradshaw Index (HBI) Disease not active: <4 ; Mild disease activity: HBI >= 4 and <= 8 ; Moderate disease activity: HBI > 8 and <= 12 ; Severe disease activity: HBI > 12
Harvey-Bradshaw Index (HBI) | Month 12
  Harvey-Bradshaw Index (HBI) Disease not active: <4 ; Mild disease activity: HBI >= 4 and <= 8 ; Moderate disease activity: HBI > 8 and <= 12 ; Severe disease activity: HBI > 12
Harvey-Bradshaw Index (HBI) | Month 18
  Harvey-Bradshaw Index (HBI) Disease not active: <4 ; Mild disease activity: HBI >= 4 and <= 8 ; Moderate disease activity: HBI > 8 and <= 12 ; Severe disease activity: HBI > 12
Harvey-Bradshaw Index (HBI) | Month 24
  Harvey-Bradshaw Index (HBI) Disease not active: <4 ; Mild disease activity: HBI >= 4 and <= 8 ; Moderate disease activity: HBI > 8 and <= 12 ; Severe disease activity: HBI > 12
Crohn's Disease Activity Index (CDAI) clinical scores | Month 6
  Crohn's Disease Activity Index (CDAI) clinical scores The patients with CD can be divided into asymptomatic remission (CDAI < 150), mild-to-moderate CD (150-220), moderate-to-severe CD (220-450), and severe-fulminant disease (>450).
Crohn's Disease Activity Index (CDAI) clinical scores | Month12
  Crohn's Disease Activity Index (CDAI) clinical scores The patients with CD can be divided into asymptomatic remission (CDAI < 150), mild-to-moderate CD (150-220), moderate-to-severe CD (220-450), and severe-fulminant disease (>450).
Crohn's Disease Activity Index (CDAI) clinical scores | Month18
  Crohn's Disease Activity Index (CDAI) clinical scores The patients with CD can be divided into asymptomatic remission (CDAI < 150), mild-to-moderate CD (150-220), moderate-to-severe CD (220-450), and severe-fulminant disease (>450).
Crohn's Disease Activity Index (CDAI) clinical scores | Month24
  Crohn's Disease Activity Index (CDAI) clinical scores The patients with CD can be divided into asymptomatic remission (CDAI < 150), mild-to-moderate CD (150-220), moderate-to-severe CD (220-450), and severe-fulminant disease (>450).
Fecal calprotectin | Month 6
  Fecal calprotectin
Fecal calprotectin | Month 12
  Fecal calprotectin

CONTACTS AND LOCATIONS:
Locations (15):
- France (15):
  - CHu de Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - CHU de Grenoble, Grenoble
  - CHU de Lille Hopital Claude Huriez, Lille
  - HCL-Hôpital Lyon Sud, Lyon
  - AP-HM Hôpital Nord, Marseille
  - CHU de Nançy, Nancy
  - CHU de Nantes, Nantes
  - Ap-HP Hopital St Louis, Paris
  - AP-HP Hôpital Européen Georges Pompidou, Paris
  - AP-HP Le Kremlin-Bicetre, Paris
  - AP-HP St Antoine, Paris
  - CHU de Rennes, Rennes
  - CHU de Strasbourg HautePierre, Strasbourg
  - CHU de Toulouse, Toulouse